CLINICAL TRIAL: NCT04567160
Title: Use of the NOL Index to Compare the Intraoperative Analgesic Effect of Propofol Versus Sevoflurane After Standardized Stimulation in Patients Under General Anesthesia. The PROSEVNOL Study
Brief Title: NOL Index to Compare the Intraoperative Analgesic Effect of Propofol Versus Sevoflurane
Acronym: PROSEVNOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Professor, MD, PhD, DESAR, Chair of Research, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-2343
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Nociceptive Pain; Anesthesia
Keywords: NOL index
MeSH Terms: conditions — Nociceptive Pain | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Active Comparator): Induction and maintenance of general anesthesia using propofol
  Interventions: Drug: Propofol
- Sevoflurane group (Active Comparator): Induction and maintenance of general anesthesia using sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — In the propofol group, general anesthesia will be induced using target-controlled infusion (TCI) of propofol and remifentanil. Marsh pharmacokinetic model will be used to set the initial target predicted effect-site concentration of propofol at 3.0 mcg/ml in flash mode. Simultaneously, target-controlled infusion of remifentanil will be started to reach an initial target predicted effect-site concentration of 3 ng/mL using the Minto pharmacokinetic model.
  After tracheal intubation, TCI of remifentanil is paused.
  Arms: Propofol group
Drug: Sevoflurane — In the sevoflurane group, induction of general anesthesia will be carried out by spontaneous breathing through a mask while progressively opening up the dial of the sevoflurane vaporizer up to 8%. Like in the propofol group, target-controlled infusion of remifentanil is simultaneously started to reach an initial target predicted effect-site concentration of 3 ng/mL. Vaporizer is adjusted when gas equilibration reaches the patient-specific concentration 1.0 MAC of sevoflurane. After tracheal intubation, TCI of remifentanil is paused.
  Arms: Sevoflurane group

SUMMARY:
The purpose of this prospective randomized controlled study is to compare the analgesic properties of propofol and sevoflurane using variation of the NOL index and standard monitoring (Heart Rate and Mean Arterial Blood Pressure) when patients under general anaesthesia with either agents are subjected to a standardized painful stimulus (a tetanic stimulation over the ulnar nerve at 70 mA, 100 Hz for 30 seconds).

DETAILED DESCRIPTION:
This study proposes a research design that compare the analgesic properties of two commonly used agents for induction and maintenance of the hypnotic component of anesthesia: propofol versus sevoflurane. Using the NOL index to quantitatively monitor nociception, it is expected to see a difference in response to a standardized electrical and tetanic stimulus during general anesthesia maintained with either agents.

Hypothesis is that magnitude of the variation and/or the value of the NOL Index following a standardized nociceptive stimulus is lower when general anesthesia is based on propofol rather than on sevoflurane.

Induction of general anesthesia will differ depending in which group the patient belongs.

In the propofol group, general anesthesia will be induced using target-controlled infusion (TCI) of propofol and remifentanil.

In the sevoflurane group, induction of general anesthesia will be carried out by spontaneous breathing through a mask while progressively opening up the dial of the sevoflurane vaporizer up to 8%. Like in the propofol group, target-controlled infusion of remifentanil is simultaneously started to reach an initial target predicted effect-site concentration of 3 ng/mL. Vaporizer is adjusted when gas equilibration reaches the patient-specific concentration 1.0 MAC of sevoflurane.

At this point, noxious stimulation will be delayed at least 10 minutes after TCI remifentanil is paused to allow for the remifentanil to be cleared out and to ensure brain-alveolar equilibration of sevoflurane (sevoflurane group).

Measurements of the NOL Index, BIS, HR and MAP start 1 minute before applying noxious stimulus (prestimulation period). Means of the data collected during that period will constitute the basal values for NOL and HR before stimulation. After this stand-by period, electric stimulation is applied. This will consist in a standardized tetanic stimulation to the ulnar nerve of the non-dominant forearm delivered by a routine nerve stimulator at a frequency of 100 Hz and a current of 70 mA for a duration of 30 seconds. Measurements of the NOL Index, BIS, HR and MAP will continue during 3 minutes after (poststimulation period). This window of recording has to be free of any other external stimulation as it could produce noise disturbance on recorded values.

After the stimulation, all the monitors will be used to guide intraoperative administration of hypnotic agents and analgesics. Total consumption of hypnotics and opioids will be recorded for the duration of surgery. Postoperative assessment of pain and opioid consumption will be done in post anesthesia care unit as exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Age 18 years or older
* Elective surgery under general anesthesia.
* Good understanding of English or French language

Non-inclusion Criteria

* Ongoing Coronary artery disease
* Patients with non-regular sinus cardiac rhythm, implanted pacemakers, prescribed antimuscarinic agents, α2-adrenergic agonists, β1-adrenergic antagonists and antiarrhythmic agents
* Emergent surgery
* Pregnancy/lactation
* Preoperative hemodynamic disturbance
* Central nervous system disorder (neurologic/head trauma/uncontrolled epileptic seizures)
* Patient refusal
* Drug or alcohol abuse within the last 6 months
* Chronic use of psychoactive drugs
* Pre-operative chronic opioid use or chronic pain, equivalent to oxycodone 20mg per oral, per day for more than 6 weeks
* History of psychiatric diseases or psychological problems
* Allergy or intolerance to any of the study drugs

Exclusion Criteria:

* Unexpected difficult airway requesting excessive, possibly painful airway manipulations.
* Intraoperative unexpected complications requiring strong hemodynamic support (transfusions, vasopressors, inotropes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Delta NOL (no unit for the NOL index) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the variation of NOL (delta NOL) after tetanic stimulation under general anesthesia based on propofol versus sevoflurane

SECONDARY OUTCOMES:
Delta Heart Rate (beat per minute) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the variation of heart rate after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Delta Mean Arterial Blood Pressure (unit: mmHg) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the variation of mean arterial blood pressure (MABP) after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Delta BIS (no unit for BIS index) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the variation of bispectral index (BIS) after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Peak value of NOL (no unit) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the peak value of NOL after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Peak value of Heart Rate (unit: beat per minute) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the peak value of heart rate after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Peak value of Mean Arterial Blood Pressure (unit: mmHg) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the peak value of mean arterial blood pressure (MABP) after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Peak value of BIS (no unit) | From 1 minute before to 3 minutes after tetanic stimulation for each patient
  To compare the peak value of bispectral index (BIS) after tetanic stimulation under general anesthesia based on propofol versus sevoflurane
Area Under the Curve for NOL for Propofol Versus Sevoflurane (no unit) | From T0 (start stimulation) to 3 minutes after tetanic stimulation for each patient
  To compare the area under the curve between propofol and sevoflurane between the beginning of stimulation and 3 minutes after stimulation
Area Under the Curve for Heart Rate for Propofol Versus Sevoflurane (no unit) | From T0 (start stimulation) to 3 minutes after tetanic stimulation for each patient
  To compare the area under the curve between propofol and sevoflurane between the beginning of stimulation and 3 minutes after stimulation
Area Under the Curve for Mean Arterial Blood Pressure for Propofol Versus Sevoflurane (no unit) | From T0 (start stimulation) to 3 minutes after tetanic stimulation for each patient
  To compare the area under the curve between propofol and sevoflurane between the beginning of stimulation and 3 minutes after stimulation
Area Under the Curve for BIS for Propofol Versus Sevoflurane (no unit) | From T0 (start stimulation) to 3 minutes after tetanic stimulation for each patient
  To compare the area under the curve between propofol and sevoflurane between the beginning of stimulation and 3 minutes after stimulation
Total Dose of Remifentanil (unit: mcg) | Intraoperative
  Total dose of remifentanil in mcg from induction of anesthesia until tracheal extubation
Total Dose of Propofol (unit: mg) | Intraoperative
  Total dose of propofol in mg from induction of anesthesia until tracheal extubation in Propofol group
Total Dose of Sevoflurane (unit: mL) | Intraoperative
  Total dose of sevoflurane in mL from induction of anesthesia until tracheal extubation in Sevoflurane group
Total Dose of Hydromorphone in post-anesthesia care unit (PACU) (unit: mg) | From entrance in post-anesthesia care unit until post-anesthesia care unit discharge, an average of 2 hours
  Total dose of hydromorphone in mg in post-anesthesia care unit
post-anesthesia care unit (PACU) Pain Scores at Rest (scale from 0 to 10) | From entrance in post-anesthesia care unit until post-anesthesia care unit discharge, an average of 2 hours
  Pain scores on a scale from 0 to 10 at rest in post-anesthesia care unit
post-anesthesia care unit (PACU) Pain Scores during Cough (scale from 0 to 10) | From entrance in post-anesthesia care unit until post-anesthesia care unit discharge, an average of 2 hours
  Pain scores on a scale from 0 to 10 during cough effort in post-anesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No